CLINICAL TRIAL: NCT02679196
Title: An Open Label Ascending Dose Study Evaluating the Safety/Tolerability, Pharmacokinetic and Pharmacodynamic Effects of KA2237 In Patients With B Cell Lymphoma
Brief Title: The Safety, Pharmacokinetic and Pharmacodynamic Effect of KA2237 (PI3 Kinase p110β/δ Inhibitor) In B Cell Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Karus Therapeutics Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KTP-002
Record Dates: First submitted 2016-01-29; First posted 2016-02-10 (Estimated); Last update posted 2019-02-06 (Actual); Status verified 2019-02

CONDITIONS: Lymphoma, B Cell
MeSH Terms: conditions — Lymphoma, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- KA2237 (Experimental): Open label treatment with KA2237
  Interventions: Drug: KA2237

INTERVENTIONS:
Drug: KA2237 — PI3 Kinase p110β/δ inhibitor
  Other Names: PI3 Kinase p110β/δ inhibitor

SUMMARY:
Multiple ascending dose study to evaluate safety/tolerability, pharmacokinetic and pharmacodynamics effects of KA2237 (PI3 Kinase p110β/δ Inhibitor) in patients with B Cell Lymphoma and determine the maximum tolerated dose (MTD) in Part I of the study. In Part II, patients with B cell lymphoma will be treated with KA2237 at the MTD to evaluate safety and efficacy in the patient population.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years at the screening visit.
2. Has given written consent to participate in the study.
3. Has B-cell lymphoma refractory to or intolerant of established therapy known to provide clinical benefit for their condition and having received rituximab as a single agent or in combination with other therapies.
4. Disease status requirement: Measurable disease defined as the presence of ≥ 1 nodal lesion that measures ≥ 1.5 cm in a single dimension as assessed by X-ray Computed Tomography (CT) (Positron Emission Tomography (PET/CT), or magnetic resonance imaging [MRI]
5. Eastern Co-operative Oncology Group (ECOG) performance status of ≤ 2.
6. For men and women of child-bearing potential, willing to use adequate contraception

Exclusion Criteria:

1. Subject is a chronic alcoholic (intake > 35 units of alcohol (>5 bottles of wine weekly)) or drug abuser
2. Subject has any medical or psychiatric condition that, in the opinion of the Investigator, may compromise the subject's ability to participate in this study
3. Female subjects who are breastfeeding, pregnant, or plan to become pregnant during the study or within 3 months following the last dose of investigational product
4. Subjects with a current or recent history, as determined by the Investigator, of severe, progressive, and/or uncontrolled renal disease (estimated glomerular filtration rate (eGFR) <30ml/min), hepatic (Alanine transaminase (ALT) 2.5 times upper limit of normal (>2.5xULN), bilirubin > 2x ULN), hematological (absolute neutrophil count (ANC) <1.0 x 109/L, platelet count <75x109/L or requires regular platelet transfusions to maintain a platelet count ≥ 75 x 109/L , hemoglobin <9g/dL), endocrine (glycated Haemoglobin (HbA1c)>7% or random glucose >200mg/dL), pulmonary (Forced Expiratory Volume in 1 second (FEV1) <70% of predicted value), cardiac (New York Heart Association (NYHA)) class III/IV, or neurological disease
5. Has had an allogeneic stem cell transplant with current active graft-versus-host-disease.
6. Has known active central nervous system involvement of the malignancy.
7. Has active, serious infection requiring systemic therapy. Patients may receive prophylactic antibiotics and antiviral therapy at the discretion of the treating physician.
8. Has a positive test for human immunodeficiency virus (HIV) antibodies.
9. Has active hepatitis B or C. Patients with serologic evidence of prior exposure are eligible.
10. Disease-related exclusions

    * Had treatment with a short course of corticosteroids (> 10mg daily prednisone equivalents) for symptom relief within 1-week prior to screening.
    * Has poorly controlled diabetes mellitus (HbA1c >7% or random glucose >200mg/dL)
    * Known tuberculosis (TB) disease or latent TB infection
    * Has chronic, active colitis
11. Medication related exclusions

    * Had alemtuzumab therapy within 12-weeks prior to screening.
    * Has taken a medication that is a potent inhibitor or inducer of cytochrome P450 3A4 (CYP3A4) within 1-week prior to screening.
    * The subject has previously participated in this study.
    * The subject has participated or is currently participating in another study of an investigational medicine or medical device (radiotherapy, radio-immunotherapy, biological therapy, chemotherapy), within 4-weeks prior to screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2016-07; Primary Completion 2018-12-24 (Actual); Study Completion 2018-12-24 (Actual)

PRIMARY OUTCOMES:
The occurrence of dose limiting toxicity (DLT); | Day 28 of treatment
  any event with possible or probable relationship to study drug occurring up to day 28 from the start of treatment as assessed using the National Cancer Institute's Common Terminology Criteria for Adverse Events version 4.03

SECONDARY OUTCOMES:
Concentration (mg/ml) of KA2237 in serum/plasma over time (hours) | 24 weeks
Concentration (mg/ml) of KA2237 in urine over time (hours) | 24 weeks
Concentration (ng/ml) of key cytokine and intracellular signalling markers in immune cell subsets | 24 weeks
Frequency of KA2237 related adverse events and laboratory abnormalities | 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Nastoupil LJ, Neelapu SS, Davis RE, Samaniego F, Fowler NH, Westin J, Lee HJ, Wang M, Hagemeister F, Cecil ARL, Dow J, Haque K, Silva FA, Whale A, Lensun L, Bone EA, McElwaine-Johnn H, Beer PA. Preclinical and phase I studies of KA2237, a selective and potent inhibitor of PI3K beta/delta in relapsed refractory B cell lymphoma. Leuk Lymphoma. 2021 Dec;62(14):3452-3462. doi: 10.1080/10428194.2021.1957874. Epub 2021 Aug 9. PMID 34365878